CLINICAL TRIAL: NCT04950192
Title: The Philips (VeriSight) Intracardiac Echocardiography (ICE) Registry
Brief Title: Philips Intracardiac Echocardiography (ICE) Clinical Registry
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019_10745
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Stroke; Valve Disease, Heart; Atrial Septal Defect; Patent Foramen Ovale; Mitral Valve Disease; Tricuspid Valve Disease; Aortic Valve Disease
Keywords: ICE; Image guided therapy; Structural Heart; Electrophysiology; Intracardiac echocardiography; Atrial Fibrillation; Stroke; Ablation; Valve Disease
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Heart Valve Diseases; Heart Septal Defects, Atrial; Foramen Ovale, Patent; Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Prospective Observational: Prospective observational subjects undergoing planned cardiac procedures utilizing image guidance
  Interventions: Device: ICE Image guidance

INTERVENTIONS:
Device: ICE Image guidance — ICE image guidance will be used on all patients undergoing planned cardiac catheterization procedures
  Other Names: Philips VeriSight ICE Catheter

SUMMARY:
The purpose of this observational registry is to report real-world safety and performance of VeriSight for ultrasound guided ICE imaging in percutaneous cardiac intervention procedures when used in standard clinical practice.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational, single-arm registry intended to gather real-world data to report VeriSight ICE catheter performance and safety. It will be conducted in the United States under the approval of one or more recognized institutional review boards and in compliance with Good Clinical Practice guidelines defined in International Standards Organization:14155;2011, the Declaration of Helsinki, and all applicable federal and local laws and regulations. Only on label uses of the VeriSight ICE catheter will be allowed. No specific claims are being validated during this registry, though data analyzed from this protocol are intended to inform of future claims regarding the performance and safety of the VeriSight catheter.

Enrolled patients will be imaged with VeriSight for various types of percutaneous cardiac interventional procedures. Enrolled subjects will be followed until discharge or ≤48 hrs post-procedure. The registry has a planned duration of approximately 24-36 months with interim analysis planned at 100 patients before further enrollment will be considered. Statistical hypotheses are not intended for this registry and descriptive analysis will be conducted. Data from all clinical sites are intended to be pooled for analysis. It is possible that sub-analyses may be conducted to demonstrate VeriSight guidance for target intervention types in structural heart and electrophysiology procedures.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and willing to provide written, dated and signed, informed consent
2. Scheduled for a procedure that is within the scope of clinical indication for VeriSight per Instructions for Use (IFU)

Exclusion Criteria:

1. Contraindicated for ICE catheter placement or patient considerations that make placement of VeriSight not technically feasible
2. If alternate access (as needed instead of femoral) is not viable
3. Known contraindicated conditions include sepsis, major coagulation abnormalities, presence of any intracardiac thrombus, presence of class IV angina or heart failure, deep vein thrombosis, or significant peripheral vascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects age 18 and older that are scheduled for and will undergo a planned cardiac interventional percutaneous procedure in which the guidance of ICE is indicated, eligible and willing to sign an informed consent without meeting any of the exclusion criteria set and meeting all the inclusion criteria set forth in the protocol will be included in the population for analyses.
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Ram, PhD, Study Director — Philips Clinical and Medical Affairs
Locations (5):
- United States (5):
  - University of Colorado, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective Observational
Started | 155
Completed | 155
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prospective Observational
Number analyzed (Participants) | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 125
  Unknown or Not Reported | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 112
  More than one race | 3
  Unknown or Not Reported | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 155

OUTCOME MEASURES:

1. Primary Outcome: Technical Success
Description: Investigator's assessment (Y/N) on successful delivery of VeriSight to the target intracardiac position and sustained device operation during the procedure
Time Frame: During procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Observational
Number analyzed (Participants) | 155
Participants | 153

2. Primary Outcome: Imaging Success
Description: Adequate image quality via Likert scale ( Acceptable or better) as determined by the investigator
Time Frame: During procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Observational
Number analyzed (Participants) | 155
Participants | 147

3. Primary Outcome: Clinical Success
Description: Investigator's assessment (Y/N) on adequacy of VeriSight imaging for visualization of major cardiac structures, and guiding procedural intervention, and ability to detect/ assess intra-procedural complications.
Time Frame: During procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Observational
Number analyzed (Participants) | 155
Participants | 149

4. Primary Outcome: Number of Participants With Device-related Adverse Event Detection
Description: Detect device-related adverse events periprocedural through discharge or ≤48 hours post-procedure, whichever is earlier.
Time Frame: Procedure through 48 hours or discharge, whichever is earlier
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective Observational
Number analyzed (Participants) | 155
Participants | 0

ADVERSE EVENTS:
Time Frame: Each subject's adverse event data were collected up to discharge or within 48 hours post procedure
Description: Adverse event reporting does not differ from clinicaltrials.gov
Arm/Group | Prospective Observational
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 0/155
Other Adverse Events (participants affected / at risk) | 0/155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or presentation concerning a single site experience may be permitted until the multi-center study has been published. Notwithstanding the foregoing or in the event such multicenter publication is not submitted within twelve (12) months of completion of the Study at all sites or if Sponsor confirms there will be no multicenter publication, Principal Investigator shall furnish Sponsor with a copy of any proposed publication or presentation at least forty-five (45) days

DOCUMENTS (2):
  • Study Protocol (2021-04-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT04950192/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT04950192/SAP_001.pdf